CLINICAL TRIAL: NCT03853291
Title: Developing a Pain Identification and Communication Toolkit for Family Caregivers of Persons With Dementia
Brief Title: Developing a Pain Identification and Communication Toolkit
Acronym: PICT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: terminated due to Covid and end of funding period for key personnel
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Cornell University (Other); Rutgers University (Other); University of Iowa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 1811019718; 3P30AG022845-15S1 (NIH)
Record Dates: First submitted 2019-02-22; First posted 2019-02-25 (Actual); Results first posted 2022-06-07 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Dementia; Chronic Pain
MeSH Terms: conditions — Dementia; Chronic Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- PICT Workbook (Experimental): PICT Workbook components includes: a) training using an observational assessment tool to detect pain in PWD, b) coaching and feedback by a research nurse in effective strategies for communicating with providers about PWD's pain, c) future planning for what steps to take when a pain symptom is detected, and d) updating the caregiver's skill set through routine practice.
  Interventions: Behavioral: PICT Workbook
- Information Pamphlet (Active Comparator): Informational pamphlet about pain in dementia and a link to the Alzheimer's Association website.
  Interventions: Behavioral: Information Pamphlet
- Family Caregivers - Interview Phase (No Intervention): Interviews will be conducted with family caregivers and health care providers in-person in private offices at WCMC/NYP or over the telephone. The primary objectives of the qualitative interviews are to: a) adapt the PAINAD for use with caregivers by asking them to comment on its format and content; and b) generate an initial question pool for the Question Prompt List. After reviewing the PICT workbook, caregivers will complete a brief qualitative questionnaire about the content, format, and perceived utility of PICT, as well as ways to enhance its cultural relevance. They will also complete a semi-structured interview to clarify their perspectives. Health care providers will answer a similar set of questions. Results from this first field-test will inform the next version of PICT and address key issues, such as the feasibility of using research nurses to administer the intervention, anticipation of participant burden for caregivers, and adequacy of PICT format and instructions.
- Healthcare Providers - Interview Phase (No Intervention): Interviews will be conducted with family caregivers and health care providers in-person in private offices at WCMC/NYP or over the telephone. The primary objectives of the qualitative interviews are to: a) adapt the PAINAD for use with caregivers by asking them to comment on its format and content; and b) generate an initial question pool for the Question Prompt List. After reviewing the PICT workbook, caregivers will complete a brief qualitative questionnaire about the content, format, and perceived utility of PICT, as well as ways to enhance its cultural relevance. They will also complete a semi-structured interview to clarify their perspectives. Health care providers will answer a similar set of questions. Results from this first field-test will inform the next version of PICT and address key issues, such as the feasibility of using research nurses to administer the intervention, anticipation of participant burden for caregivers, and adequacy of PICT format and instructions.
- Family Caregivers - Field Test Phase (No Intervention): Once initial versions of the PICT manual and workbook are developed, they will be iteratively field-tested and vetted by family caregivers and health care providers. After reviewing the PICT workbook, caregivers will complete a brief qualitative questionnaire about the content, format, and perceived utility of PICT, as well as ways to enhance its cultural relevance. They will also complete a brief (15-20 minute) semi-structured interview to clarify their perspectives. Health care providers will answer a similar set of questions. Results from this first field-test will inform the modified version of PICT and will address key issues, such as the feasibility of using research nurses (and other practice staff) to administer the intervention, anticipation of participant burden for caregivers, and adequacy of PICT format and instructions.
- Healthcare Providers - Field Test Phase (No Intervention): Once initial versions of the PICT manual and workbook are developed, they will be iteratively field-tested and vetted by family caregivers and health care providers. After reviewing the PICT workbook, caregivers will complete a brief qualitative questionnaire about the content, format, and perceived utility of PICT, as well as ways to enhance its cultural relevance. They will also complete a brief (15-20 minute) semi-structured interview to clarify their perspectives. Health care providers will answer a similar set of questions. Results from this first field-test will inform the modified version of PICT and will address key issues, such as the feasibility of using research nurses (and other practice staff) to administer the intervention, anticipation of participant burden for caregivers, and adequacy of PICT format and instructions.

INTERVENTIONS:
Behavioral: PICT Workbook — PICT Workbook: The PICT workbook is a 31-page manual, which includes: a) training using an observational assessment tool to detect pain in PWD, b) coaching and feedback by a research nurse in effective strategies for communicating with providers about PWD's pain, c) future planning for what steps to take when a pain symptom is detected, and d) updating the caregiver's skill set. Participants in the intervention condition also attended four weekly 30-minute sessions with an interventionist through a combination of online (video observation) and telephone coaching to go over the Workbook.
  Arms: PICT Workbook
Behavioral: Information Pamphlet — Pamphlet with information about pain and dementia and links to Alzheimer's Association
  Arms: Information Pamphlet

SUMMARY:
The proposed research will develop, refine, and pilot test the Pain Identification and Communication Toolkit (PICT), an intervention to help family caregivers of community-dwelling persons with dementia identify pain symptoms and communicate those symptoms to health care providers. Informed by self-efficacy theory, PICT will include: a) training in administering an observational assessment tool to identify pain in persons with dementia, b) coaching in effective communication about the person with dementia's pain symptoms, c) future planning for steps to take when pain is detected, and d) updating caregivers' skills through routine practice with the pain assessment tool. All components will be vetted and iteratively field-tested with a sample of racially and ethnically diverse caregivers of community-dwelling persons with dementia and health care providers. A two-group pilot randomized trial will examine the acceptability, feasibility, and preliminary impact of PICT on caregivers' initiation of pain-related communication with health care providers.

ELIGIBILITY:
For all phases:

Inclusion Criteria:

* Family caregiver
* Age 21 or older
* English speaking
* Cognitively intact
* Provides at least 8 hours of care per week to a person with dementia and pain
* Has provided care for at least 6 months

Exclusion Criteria:

* Paid caregiver
* Age 20 or younger
* Non-English speaking
* Cognitively impaired
* Does not provide at least 8 hours of care per week to a person with dementia who also has a pain diagnosis
* Has not provided care for at least 6 months
* Currently enrolled in hospice
* The patient to whom the caregiver provides assistance is in enrolled in hospice
* Care recipient does not have dementia diagnosis or pain diagnosis

For field test and interview phases:

Healthcare professionals:

* Currently providing clinical services to persons with dementia and/or chronic pain
* Has provided these clinical services for at least 1 year

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2019-03-08 (Actual); Primary Completion 2021-08-11 (Actual); Study Completion 2021-08-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cary Reid, MD/PhD, Principal Investigator — Weill Medical College of Cornell University; Catherine Riffin, PhD, Principal Investigator — Weill Medical College of Cornell University; Karl Pillemer, PhD, Principal Investigator — Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Riffin C, Brody L, Mukhi P, Herr K, Pillemer K, Rogers M, Henderson CR Jr, Reid MC. Establishing the Feasibility and Acceptability of a Caregiver Targeted Intervention to Improve Pain Assessment Among Persons With Dementia. Innov Aging. 2023 Jul 13;7(10):igad074. doi: 10.1093/geroni/igad074. eCollection 2023. PMID 38094933

RESULTS

PARTICIPANT FLOW:
Groups:
- PICT Workbook: PICT Workbook: The PICT workbook is a 31 page manual, which includes: a) training using an observational assessment tool to detect pain in PWD, b) coaching and feedback by a research nurse in effective strategies for communicating with providers about PWD's pain, c) future planning for what steps to take when a pain symptom is detected, and d) updating the caregiver's skill set. Participants in the intervention condition also attended four weekly 30-minute sessions with an interventionist through a combination of online (video observation) and telephone coaching to go over the Workbook.
Period: Overall Study
Arm/Group | PICT Workbook | Information Pamphlet | Family Caregivers - Interview Phase | Healthcare Providers - Interview Phase | Family Caregivers - Field Test Phase | Healthcare Providers - Field Test Phase
Started | 18 | 16 | 18 | 16 | 6 | 11
Completed | 16 | 13 | 18 | 16 | 6 | 11
Not Completed | 2 | 3 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 2 | 0 | 0 | 0 | 0
Not completed — Determined to be ineligible | 1 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PICT Workbook | Information Pamphlet | Family Caregivers - Interview Phase | Healthcare Providers - Interview Phase | Family Caregivers - Field Test Phase | Healthcare Providers - Field Test Phase | Total
Number analyzed (Participants) | 18 | 16 | 18 | 16 | 6 | 11 | 85
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Age was not collected from healthcare providers
  years
    number analyzed (Participants) | 18 | 16 | 18 | 0 | 6 | 0 | 58
    (all) | 63.1 (9.72) | 61.6 (9.14) | 61.5 (11.63) |  | 61.67 (9.35) |  | 62.0 (9.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 16 | 15 | 12 | 6 | 8 | 72
  Male | 3 | 0 | 3 | 4 | 0 | 3 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 3 | 1 | 1 | 1 | 10
  Not Hispanic or Latino | 15 | 14 | 15 | 14 | 5 | 10 | 73
  Unknown or Not Reported | 1 | 0 | 0 | 1 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 2 | 5 | 0 | 2 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Black or African American | 3 | 2 | 3 | 0 | 0 | 0 | 8
  White | 12 | 11 | 12 | 10 | 6 | 8 | 59
  More than one race | 2 | 1 | 1 | 0 | 0 | 0 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 18 | 16 | 18 | 16 | 6 | 11 | 85

OUTCOME MEASURES:

1. Primary Outcome: Feasibility, as Measured by the Number of Participants in the Intervention Condition Who Completed All Sessions
Time Frame: Post-intervention, 3 months
Population: 2 participants did not complete the intervention, n=1 lost to follow-up, n=1 determined ineligible post-enrollment. Data were not collected from participants in the interview and field test arms/phases.
Measure: Count of Participants; unit: Participants
Arm/Group | PICT Workbook
Number analyzed (Participants) | 16
Participants | 16

2. Primary Outcome: Feasibility, as Measured by the Number of Participants Recruited
Time Frame: Baseline
Population: Data were not collected from participants in the interview and field test arms/phases.
Measure: Count of Participants; unit: Participants
Arm/Group | PICT Workbook | Information Pamphlet
Number analyzed (Participants) | 18 | 16
Participants | 18 | 16

3. Primary Outcome: Acceptability, as Measured by the Number of Participants Who Report That the Intervention Was "Very Effective" or "Moderately Effective" in Helping Them Feel More Confident in Their Ability to Communicate Pain to Healthcare Providers
Time Frame: Post-intervention, 3 months
Population: For the intervention condition: 2 participants did not complete the intervention, n=1 lost to follow-up, n=1 determined ineligible post-enrollment. Data from the information pamphlet arm was not collected. Data were not collected from participants in the interview and field test arms/phases.
Measure: Count of Participants; unit: Participants
Arm/Group | PICT Workbook
Number analyzed (Participants) | 16
Participants | 13

4. Secondary Outcome: Caregiver Initiated Pain-related Communication, as Measured by the Number of Caregivers Who Report Making Contact With Any of the Care Recipients' Health Care Providers to Discuss Pain-related Concerns
Time Frame: Baseline, Post-intervention-3 months
Population: 5 participants overall were not analyzed. For the workbook: n=1 lost to follow-up, n=1 deemed ineligible. For informational pamphlet: n=2 lost to follow-up, n=1 deemed ineligible. Data were not collected from participants in the interview and field test arms/phases.
Measure: Count of Participants; unit: Participants
Groups:
- Informational Pamphlet: Informational pamphlet about pain in dementia and a link to the Alzheimer's Association website.
  Information Pamphlet: Pamphlet with information about pain and dementia and links to Alzheimer's Association
Arm/Group | PICT Workbook | Informational Pamphlet
Number analyzed (Participants) | 16 | 13
Participants
  Baseline | 13 | 8
  3 Month Assessment | 12 | 8

ADVERSE EVENTS:
Time Frame: Up to 3 months.
Description: Participants were assessed for SAEs and safety alerts. SAEs included caregiver hospitalization, institutionalization, ER visit, and death. Safety alerts included severe medical problem of the caregiver, caregiver or care recipient abuse, caregiver threatens to harm themselves or disruptions in caregiver/patient relationship. Safety alerts were not considered SAEs. All-Cause Mortality, Serious, and Other AE data were not collected for "Interview Phase" and the "Field Test Phase" Arms/Groups.
Groups:
- PICT: Pain Identification and Communication Toolkit (PICT) components include: a) training using an observational assessment tool to detect pain in persons with dementia, b) coaching and feedback by a research nurse in effective strategies for communicating with providers about their care recipient's pain, c) future planning for what steps to take when a pain symptom is detected, and d) updating the caregiver's skill set through routine practice.
  PICT: PICT is a manualized, multicomponent intervention delivered by a trained interventionist. PICT consists of 4 weekly telephone sessions (30-60 mins each) guided by an Instructor Manual and companion Caregiver Workbook
- Control Group: Informational pamphlet about pain in dementia and a link to the Alzheimer's Association website.
  Information Pamphlet: Pamphlet with information about pain and dementia and links to Alzheimer's Association
Arm/Group | PICT | Control Group | Family Caregivers - Interview Phase | Healthcare Providers - Interview Phase | Family Caregivers - Field Test Phase | Healthcare Providers - Field Test Phase
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/16 | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/16 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/18 | 0/16 | 0/0 | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
This is a pilot RCT focused on feasibility and acceptability, and was not fully powered to evaluate the intervention's efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-17): https://cdn.clinicaltrials.gov/large-docs/91/NCT03853291/Prot_SAP_000.pdf